CLINICAL TRIAL: NCT02683759
Title: The Efficacy and Tolerability of Bio-Enhanced Curcumin in Maintaining Remission in Patients With Ulcerative Colitis
Brief Title: Bio-enhanced Curcumin as an Add-on Treatment in Maintaining Remission of Ulcerative Colitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Rupa Banerjee, Consultant Gastroenterologisy, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AIGINDIACurcumin2
Record Dates: First submitted 2016-02-10; First posted 2016-02-17 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Arm (Active Comparator): Patients will receive 5-Aminosalicyclic acid as per their current treatment regimen and will also take Bio-enhanced curcumin twice daily after meals as per the following regimen:
  Interventions: Dietary Supplement: Bio-enhanced Curcumin Soft Gelatin Capsule; Drug: 5-Aminosalicyclic acid
- Control Arm (Placebo Comparator): Patients will receive 5-Aminosalicyclic acid as per their current treatment regimen and will also take a placebo pill twice daily after meals
  Interventions: Drug: 5-Aminosalicyclic acid

INTERVENTIONS:
Dietary Supplement: Bio-enhanced Curcumin Soft Gelatin Capsule — Each capsule is a bio-enhanced modification of curcumin (diferuloylmethane), which is a derivative of curcuma longa (rhizome extract)
  Starting dose: 50 mg BID of Bioenhanced Curcumin Increase dose to 100 mg BID after two (2) weeks if there is no response to the drug
  Other Names: Valdone
  Arms: Treatment Arm
Drug: 5-Aminosalicyclic acid — Dosage is as instructed by patient's physician
  Other Names: 5-ASA

SUMMARY:
Inflammatory Bowel Disease, including ulcerative colitis, is thought to result from an imbalance of pro-inflammatory and anti-inflammatory factors. As such, the majority of treatment options are directed at attempting to control the chronic inflammation and prolonging remission of clinical symptoms. Several studies have proven that curcumin has well-established anti-inflammatory properties. However, curcumin has poor bioavailability and prior studies have needed to use high concentrations in order to study the efficacy of the product. The investigators propose that a bio-enhanced preparation of curcumin will require a lower dosage to reach and affect its target tissue and will subsequently produce less adverse side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been in symptomatic remission from Ulcerative Colitis for at least 3 months. This is defined as a Partial Mayo Index Score of 0 or 1
* Age 18 years and above
* Male or female
* Patients who are able and willing to follow the treatment given and record responses in survey form

Exclusion Criteria:

* Patients who are currently experiencing symptomatic flares of mild or moderate ulcerative colitis, or have a partial mayo index score of 2 or greater
* Patients who have been taking azathioprine or mercaptopurine for <12 weeks for the treatment of their ulcerative colitis
* Patients who are taking steroids, immunosuppressants, or biologic agents for the treatment of their ulcerative colitis
* Patients who have severe ulcerative colitis
* Patients who are noncompliant with medication or regular follow up visits
* Patients who are unable or unwilling to record their responses in survey form
* Patients with comorbid illnesses, including: Diabetes Mellitus, Stage III or above Congestive Heart Failure, chronic pancreatitis, severe liver or renal disease
* Patients who have current gallstones or biliary dysfunction
* Patients with anemia (Hemoglobin <10), thrombocytopenia, abnormal lymphocyte counts, or coagulation abnormalities
* Patients with current sepsis or current ongoing infection, including C. difficile colitis or enteritis
* Patients with a history of malignancy
* Patients who are currently pregnant or nursing
* Patients who are current smokers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who remained in clinical remission in the treatment arm compared with percentage of patients who remained in clinical remission in the control arm | 1 year
  Clinical remission is recorded by a Partial Mayo Index score of 0-1
Percentage of patients who remained in endoscopic remission in the treatment arm compared with percentage of patients who remained in endoscopic remission in the control arm | 1 year
  Endoscopic remission is defined as endoscopic mucosal healing, is recorded by a Ulcerative Colitis Endoscopic Index of Severity (UCEIS) score of <3

SECONDARY OUTCOMES:
Percentage of patients in the treatment arm who experienced adverse events as compared with patients in the placebo arm | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rupa Banerjee, MD, DM, Principal Investigator — Asian Institute of Gastroenterology
Locations (1):
- Asian Institutes of Gastroenterology, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No